CLINICAL TRIAL: NCT05687396
Title: Virtual Reality in Chronic Obstructive Pulmonary Disease: Randomized Contolled Trial
Brief Title: Virtual Reality in COPD Exacerbation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Erhan KIZMAZ, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Doktora
Record Dates: First submitted 2022-12-25; First posted 2023-01-18 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: COPD Exacerbation; Pulmonary Rehabilitation
Keywords: COPD, pulmonary rehabilitation, virtual reality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual reality (Experimental): Virtual reality while cycling with ergometer in addition to conventional pulmonary rehabilitation. virtual reality designed as cylcling in the forest.
  Interventions: Device: virtual reality
- Conventional pulmonary rehabilitation (Experimental): Deep diafragmatic breathing exercise, chest expansion exercies, pursed lip exhalation, coughing and huffing, upper limp exercies with deep breathing exercise, standing up-right position, cycling with ergometer.
  Interventions: Other: conventional pulmonary rehabilitation

INTERVENTIONS:
Device: virtual reality — virtual reality designed as cycling in the forest
  Arms: Virtual reality
Other: conventional pulmonary rehabilitation — pulmonary rehabilitation
  Arms: Conventional pulmonary rehabilitation

SUMMARY:
In addition to conventional pulmonary rehabilitation, virtual reality will be applied during the hospitalization period of individuals hospitalized for COPD exacerbation. It is aimed to get more efficiency from the interventions in this short time.

DETAILED DESCRIPTION:
Subjects with COPD exacerbation will be divided two groups. Group-1 will exercise with a bicycle ergometer until fatigue in addition to pulmonary rehabilitation. Group-2 will do the same exercises. Subjects in Group-2 will use virtual reality simulation, which is designed as cycling in the forest while cycling. Treatment will continue until discharge. CAT score, mMRC dyspnea score, hospital anxiety and depression score and London chest daily living activity score will be examined before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are in COPD exacerbation period, FEV1 <70%, GOLD 2-3 spirometric stage, Hodkinson mental test score > 6 and who want to participate in the study voluntarily will be included in the study.

Exclusion Criteria:

* If there is respiratory disease considered more significant than COPD (bronchiectasis, lung cancer requiring active therapy, or asthma), Heart failure New York Heart Association (NYHA) stage 3-4, Significant hemoptysis, surgical or non-surgical lung volume in the past 6 months Individuals with reduction procedures, Lung transplantation or pneumonectomy surgery in the last 6 months, pulmonary embolism or pulmonary edema, acute myocardial infarction, acute heart failure, vertigo, epilepsy and visual impairment will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04-10 (Estimated); Study Completion 2024-04-22 (Estimated)

PRIMARY OUTCOMES:
1 minute sit and stand test | 5 minutes
  performance
Chronic Obstructive Pulmonary Disease Assessment Test | 3-7 days
  The test assessts COPD symptoms, higher scores mean bad stiation
London chest activity of daily living | 3-7 days
  The test assessts dyspnea that occurs during daily living activities. The total score can range from 0 to 75 points, with higher values translating to greater limitation in activities of daily living.
Hospital anxiety and depression scale | 3-7 days
  The test has 2 subparameter as anxiety and depression. Each question in the test contains 4 options expressing frequency on a scale 0 to 3. Higher scores mean bad stiation for each parameter.
Modified Medical Research Council | 3-7 days
  The test has 5 options thas describe dyspnea. Higher scores mean higher dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan Kızmaz, Msc, Principal Investigator — Pamukkale University; Orçin Telli Atalay, professor, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Pamukkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kizmaz E, Telli Atalay O, Cetin N, Ugurlu E. Virtual reality for COPD exacerbation: A randomized controlled trial. Respir Med. 2024 Aug-Sep;230:107696. doi: 10.1016/j.rmed.2024.107696. Epub 2024 Jun 8. PMID 38857811